CLINICAL TRIAL: NCT05363462
Title: Use of Topical Broad-spectrum Antibiotics as a Prophylaxis for Surgical Site Infection
Brief Title: Topical Antibiotics in Surgical Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OR20-00007
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Surgical Site Infection; Complication of Surgical Procedure
Keywords: Antibiotic; Surgical site infection; Ankle fractures; Complication
MeSH Terms: conditions — Surgical Wound Infection; Ankle Fractures | interventions — Vancomycin; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Two groups of treatment with a surgical ankle fracture
  1. Surgical treatment
  2. Surgical treatment plus 1 g of topical vancomycin
Who Masked: Participant
Masking Description: The patients involved in the protocol will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ankle fracture surgical treated plus 1 g of topical vancomycin (Experimental): A standard surgical treatment of patients with ankle fracture must be carried out. Classified according to Danis Webber classification system. Plus application of 1 g of vancomycin in powder in the surgical site
  Interventions: Drug: Vancomycin 1000 MG
- Ankle fracture surgical treated (Active Comparator): A standard surgical treatment of patients with ankle fracture must be carried out. Classified according to Danis Webber classification system
  Interventions: Drug: Vancomycin 1000 MG

INTERVENTIONS:
Drug: Vancomycin 1000 MG — Application of vancomycin in powder in the surgical site of treatment before closure of surgical wound
  Other Names: antibiotic; vancomycin

SUMMARY:
Ankle fractures are one of the most common injuries in traumatology. It is the fourth most common fracture in general population after hip, wrist, and hand fractures. These injuries are the second cause of hospitalization due to fractures.

Surgical site infections can be divided according to the Center of Disease Control (CDC) in superficial surgical site infections whose are defined as any infection that happens within the next 30 days after the procedure, they involve only the skin and subcutaneous tissue of the incision, and the patient presents at least one of the following: purulent drainage of the superficial incision, microorganisms isolation from an aseptically obtained culture of body fluid or tissue or the pain existence, tenderness or local inflammation at the superficial incision site despite negative cultures. Also, a diagnosis made by the surgeon or attending medic.

DETAILED DESCRIPTION:
Ankle fractures are one of the most common injuries in traumatology. It is the fourth most common fracture in general population after hip, wrist, and hand fractures. These injuries are the second cause of hospitalization due to fractures. Despite the improvement in the ankle fracture management, it has been estimated that the ankle fracture incidence has been increasing and one of the motives is an increase of ageing population. It has been estimated that ankle fractures have an incidence between 71 to 187 cases per 100,000 inhabitants a year.

Most of the ankle fractures are due to fallings or traffic accidents, it has been reported that up to 71% from ankle fracture causes are due to mechanisms of low energy, especially among the elderly and those with comorbidities these injuries are commonly caused by the inversion of the ankle, where the force and weight of the body falls in the fibula, which in young individuals usually results in only an ankle sprain, being the conservative management the most effective treatment. Nevertheless, in aging patients, these same mechanisms can provoke a fracture.

Ankle fractures represent a challenge for the orthopedic surgeon because in this very joint, despite being relatively stable, rests the entire bodyweight and a correct approach is required for the functionality to not being affected.

Ankle fractures are classified according to AO/OTA and Danis-Weber classifications. Single malleolus fractures are the most frequent (43.7 - 10%) and inside the Orthopedic Trauma Association (OTA) classification, type B are more common with a 65.8%, which tend to be displaced fractures. In patients with unstable or displaced fractures, or where a severe dislocation exists, surgical intervention is advised.

These injuries require a surgical treatment, which brings another issue: surgical site infections.

Surgical site infections can be divided according to the CDC in superficial surgical site infections whose are defined as any infection that happens within the next 30 days after the procedure, they involve only the skin and subcutaneous tissue of the incision, and the patient presents at least one of the following: purulent drainage of the superficial incision, microorganisms isolation from an aseptically obtained culture of body fluid or tissue or the pain existence, tenderness or local inflammation at the superficial incision site despite negative cultures. Also, a diagnosis made by the surgeon or attending medic.

Deep incisional surgical site infections are defined as:

1. An infection that occurs within the next 30 days after the surgery if no implant is there or a year after the surgery if there is an implant and the infection seems to be related with the procedure, where involves the deep tissue as fascial and muscular layers and presents:

   1. Purulent drainage from the deep incision
   2. Surgical incision that opens spontaneously or deliberately opened by a surgeon, and a positive culture
2. If there is no positive culture, the presence of fever (> 38° Celsius degrees), pain or tenderness.
3. An abscess or a diagnosis made by a surgeon or the attending medic. There are established risk factors for the development of surgical site infections, some of them are patient age, nutritional state, diabetes, smoking, obesity, altered immune state (8) and bacteria colonization due to contamination. This is relevant because S. aureus, negative coagulase Staphylococcus or Enterococcus are the most common causal agents for surgical site infections, which tend to be multiresistant to the most used antibiotics.

There is controversy in the prophylactic usage of antibiotics in the management of surgical injuries. The available literature supports the usage of prophylactic IV antibiotics 1 hour prior procedure and until 48 hours after, as defined by lead surgeon. Other prophylactic management is the usage of topical broad-spectrum antibiotics.

The information about the usage of topical broad-spectrum antibiotics is equally controversial. Topical vancomycin is advised in patients with surgeries that involve a high risk of developing severe and resistant infections such as spine, thorax, or cranium surgery, where its application has shown a decrease of surgical site infection acquisition risk. In one study, topical antibiotic application was carried out by irrigating 2.5 g of Vancomycin dissolved in 2 mL of saline solution before sternum incision, and at the procedure ending after injury closure. In some other studies 1 g of Vancomycin powder was placed over the cranium, then irrigated with saline solution before injury closure.

Nevertheless, these prophylaxis therapy has not been evaluated in patients under open ankle surgery with intern fixation. The available literature about these patients' management doesn´t oppose to the general surgical site infection guidelines.

ELIGIBILITY:
Inclusion Criteria:

* • Patients older than 18 years

  * Patients with a closed fracture independently of mechanism and classification
  * Patients who require an open reduction with internal fixation surgery
  * Patients who decide to participate in the study

Exclusion Criteria:

* Patients with exposed fractures
* Presence of any form of immune deficiency
* Vancomycin hyper sensibility
* Surgery in the affected ankle within the last six months
* Steroid usage
* Antibiotic usage one week prior entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Rate of surgical infection site | 90 days
  Defined as the number of patients with surgical infection site from the total of evaluated patients included in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario "Dr. José E. González", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Juto H, Nilsson H, Morberg P. Epidemiology of Adult Ankle Fractures: 1756 cases identified in Norrbotten County during 2009-2013 and classified according to AO/OTA. BMC Musculoskelet Disord. 2018 Dec 13;19(1):441. doi: 10.1186/s12891-018-2326-x. PMID 30545314
- [Result] Goost H, Wimmer MD, Barg A, Kabir K, Valderrabano V, Burger C. Fractures of the ankle joint: investigation and treatment options. Dtsch Arztebl Int. 2014 May 23;111(21):377-88. doi: 10.3238/arztebl.2014.0377. PMID 24939377
- [Result] Sun Y, Wang H, Tang Y, Zhao H, Qin S, Xu L, Xia Z, Zhang F. Incidence and risk factors for surgical site infection after open reduction and internal fixation of ankle fracture: A retrospective multicenter study. Medicine (Baltimore). 2018 Feb;97(7):e9901. doi: 10.1097/MD.0000000000009901. PMID 29443762
- [Result] Golano P, Vega J, de Leeuw PA, Malagelada F, Manzanares MC, Gotzens V, van Dijk CN. Anatomy of the ankle ligaments: a pictorial essay. Knee Surg Sports Traumatol Arthrosc. 2010 May;18(5):557-69. doi: 10.1007/s00167-010-1100-x. Epub 2010 Mar 23. PMID 20309522
- [Result] Elsoe R, Ostgaard SE, Larsen P. Population-based epidemiology of 9767 ankle fractures. Foot Ankle Surg. 2018 Feb;24(1):34-39. doi: 10.1016/j.fas.2016.11.002. Epub 2016 Nov 18. PMID 29413771
- [Result] Shao J, Zhang H, Yin B, Li J, Zhu Y, Zhang Y. Risk factors for surgical site infection following operative treatment of ankle fractures: A systematic review and meta-analysis. Int J Surg. 2018 Aug;56:124-132. doi: 10.1016/j.ijsu.2018.06.018. Epub 2018 Jun 18. PMID 29929022
- [Result] Ban KA, Minei JP, Laronga C, Harbrecht BG, Jensen EH, Fry DE, Itani KM, Dellinger EP, Ko CY, Duane TM. American College of Surgeons and Surgical Infection Society: Surgical Site Infection Guidelines, 2016 Update. J Am Coll Surg. 2017 Jan;224(1):59-74. doi: 10.1016/j.jamcollsurg.2016.10.029. Epub 2016 Nov 30. No abstract available. PMID 27915053
- [Result] Gross CE, Green CL, DeOrio JK, Easley M, Adams S, Nunley JA 2nd. Impact of Diabetes on Outcome of Total Ankle Replacement. Foot Ankle Int. 2015 Oct;36(10):1144-9. doi: 10.1177/1071100715585575. Epub 2015 May 6. PMID 25948694
- [Result] Martin ET, Kaye KS, Knott C, Nguyen H, Santarossa M, Evans R, Bertran E, Jaber L. Diabetes and Risk of Surgical Site Infection: A Systematic Review and Meta-analysis. Infect Control Hosp Epidemiol. 2016 Jan;37(1):88-99. doi: 10.1017/ice.2015.249. Epub 2015 Oct 27. PMID 26503187
- [Result] Li S, Rong H, Zhang X, Zhang Z, Wang C, Tan R, Wang Y, Zheng T, Zhu T. Meta-analysis of topical vancomycin powder for microbial profile in spinal surgical site infections. Eur Spine J. 2019 Dec;28(12):2972-2980. doi: 10.1007/s00586-019-06143-6. Epub 2019 Sep 14. PMID 31522274
- [Result] Owen MT, Keener EM, Hyde ZB, Crabtree RM, Hudson PW, Griffin RL, Lowe JA. Intraoperative Topical Antibiotics for Infection Prophylaxis in Pelvic and Acetabular Surgery. J Orthop Trauma. 2017 Nov;31(11):589-594. doi: 10.1097/BOT.0000000000000941. PMID 28708777
- [Result] Mallela AN, Abdullah KG, Brandon C, Richardson AG, Lucas TH. Topical Vancomycin Reduces Surgical-Site Infections After Craniotomy: A Prospective, Controlled Study. Neurosurgery. 2018 Oct 1;83(4):761-767. doi: 10.1093/neuros/nyx559. PMID 29267955